CLINICAL TRIAL: NCT05804344
Title: Establish the Role of Premotor and Motor Cortices in tDCS-facilitated Speech Motor Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 206731
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All five groups are compared in a linear mixed effects model.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Device is pre-set so that individual applying stimulation does not know what condition is being applied. Participants are not informed either. All data are coded by individuals who are not informed as to the condition of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Anodal speech motor tDCS (Anode: C5; Cathode: Fp2) (Experimental): Speech motor learning task performed with the stimulation condition in the arm title.
  Interventions: Device: Anodal speech motor tDCS
- Cathodal speech motor tDCS (Anode: Fp2; Cathode: C5) (Active Comparator): Speech motor learning task performed with the stimulation condition in the arm title.
  Interventions: Device: Cathodal speech motor tDCS
- Anodal IFG tDCS (Anode: F3; Cathode: Fp2) (Active Comparator): Speech motor learning task performed with the stimulation condition in the arm title.
  Interventions: Device: Anodal IFG tDCS
- Cathodal IFG tDCS (Cathode: F3; Anode: Fp2) (Active Comparator): Speech motor learning task performed with the stimulation condition in the arm title.
  Interventions: Device: Cathodal IFG tDCS
- Sham tDCS (Sham Comparator): Speech motor learning task performed with the stimulation condition in the arm title.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal speech motor tDCS — tDCS montage set for Anode: C5; Cathode: Fp2
  Arms: Anodal speech motor tDCS (Anode: C5; Cathode: Fp2)
Device: Cathodal speech motor tDCS — tDCS montage set for Anode: Fp2; Cathode: C5
  Arms: Cathodal speech motor tDCS (Anode: Fp2; Cathode: C5)
Device: Anodal IFG tDCS — tDCS montage set for Anode: F3; Cathode: Fp2
  Arms: Anodal IFG tDCS (Anode: F3; Cathode: Fp2)
Device: Cathodal IFG tDCS — tDCS montage set for Anode: Fp2; Cathode: F3
  Arms: Cathodal IFG tDCS (Cathode: F3; Anode: Fp2)
Device: Sham tDCS — tDCS device set in Sham mode
  Arms: Sham tDCS

SUMMARY:
Groups of unimpaired participants will all receive speech motor training of nonwords, and six tDCS conditions will be compared: anodal tDCS over speech motor regions; cathodal tDCS over speech motor regions; anodal tDCS over left frontal regions; cathodal tDCS over left frontal regions; cathodal stimulation over non-speech motor regions (anodal already collected);and sham tDCS (no stimulation). This will address a basic science question about whether the mechanism underlying speech motor learning requires premotor and motor cortical regions to be stimulated, which has implications for treatment of acquired speech impairment. The primary outcome measure will be the difference in production accuracy and changes in motor acuity (measured with duration) of novel consonant cluster production.

DETAILED DESCRIPTION:
Study Overview

Groups of unimpaired participants will all receive speech motor training of nonwords, and six tDCS conditions will be compared: anodal tDCS over speech motor regions; cathodal tDCS over speech motor regions; anodal tDCS over left frontal regions; cathodal tDCS over left frontal regions; cathodal stimulation over non-speech motor regions (anodal already collected);and sham tDCS (no stimulation). This will address a basic science question about whether the mechanism underlying speech motor learning requires premotor and motor cortical regions to be stimulated, which has implications for treatment of acquired speech impairment. The primary outcome measure will be the difference in production accuracy and changes in motor acuity (measured with duration) of novel consonant cluster production.

Methods & Procedures Participants will come to the testing room and the procedure will be discussed with them. This will include familiarizing them with the tDCS device and explaining how it works, ensuring once again that they do not meet any of the exclusion criteria, and explaining the possible side effects of transient tingling and/or reddening during the stimulation. We will explain that all appropriate protections are in place. We will also explain the single-blind nature of the study in that the participants may receive either active stimulation or sham stimulation. The explanation and the stimulation itself will be performed by individuals who have received training and certification in the safe use of tDCS. After determining the participant's eligibility for the study through familiarization with the equipment, they will fill out the consent form. In total, there will be two visits, with the first visit lasting approximately 85 minutes and the second visit approximately 15-20 minutes.

Speech Stimuli. The speech stimuli are disyllabic nonwords beginning with non-native native consonant clusters (e.g., GDEEVOO; FNEEGDWOP). Eight non-native clusters will be used, with four nonwords for each cluster trained during the practice session and four saved for retention session testing. All nonwords will contain legal English sounds and sequences other than the initial consonant cluster, but differ in the Consonant-Vowel (CV) shape of the syllables (e.g., GDEEVOO /gdivu/ has the shape [CCV.CV]; FNEEGDWOP /fnigdw?p/ has the shape [CCVC.CCVC]). The auditory stimuli have already been recorded by a phonetically-trained Russian-English bilingual speaker using a Shure SM-10 head-mounted microphone attached to a Marantz PMD660 digital recorder. The soundfiles were spliced to leave 10ms of silence at the onset and offset of each item using Praat, and the stimulus amplitude was normalized. Orthographic versions of the nonwords were also presented to participants to ensure that errors in cluster production did not arise from misperception.

Speech motor learning task procedure. All testing will take place in a sound-attenuated testing room. Participants will sit in front of a computer and their productions were recorded using a Shure BETA 58A microphone in a desktop microphone stand connected to the Marantz PMD660. This setup permits the participant to have the tDCS setup on their scalp throughout the learning task.

Pre-practice. To ensure that individuals understand the task, we will provide two items in pre-practice ("FTAKE" and "FNIP"). These items have been selected because English listeners' perception of these clusters is typically accurate, allowing us to easily provide accurate feedback. We will provide instructions about accurately producing consonant clusters for everyone. Pre-practice will last approximately two minutes.

Practice. During practice, participants will produce 4 nonwords per cluster (32 nonwords with illegal clusters total) seven times each along with 62 filler stimuli not containing clusters. Random stimulus presentation orders have been generated and modified to ensure that no stimulus is presented twice in succession. Items will be balanced across participants such that half of the participants will be trained on one half of the nonwords and the other half on the other nonwords. For each stimulus, participants will be presented with both auditory and orthographic versions simultaneously. The practice session will be structured to include a large amount of practice of the clusters presented randomly and in varied contexts. No online feedback will be provided given the difficulty of perceiving the accuracy of these clusters. The entire practice session will last approximately 25 minutes.

Retention. The shorter-term retention (R1) and longer-term retention (R2) sessions will be identical, with R1 beginning approximately 30 minutes after the end of practice, and R2 taking place in a separate session two days later. For each cluster, participants will produce the four trained nonwords as well as four novel, untrained nonwords beginning with the cluster. Each stimulus will be produced three times (192 total cluster stimuli) during the retention sessions, with an additional 110 filler items not containing clusters. The stimuli will be randomized and presented electronically.

tDCS procedure. The tDCS electrodes will placed on all participants in the appropriate configuration for their randomly assigned group. Participants will spend the first 10 minutes of stimulation performing computerized working memory tasks (e.g., forwards and backwards digit and block span, all with keyboard or button box responses), consistent with our previous finding that stimulation before the speech learning task can facilitate additional learning. A 1x1 Soterix battery-driven current stimulator delivered current using rubber-carbon electrodes (35cm2) with surrounding saline-soaked sponges. The electrodes will be placed based upon the randomly assigned condition with sham electrode placement split among the electrode configurations. For participants receiving active tDCS, the device will deliver 1mA of current for 20 minutes. For sham tDCS, the current will ramp up to 1mA over 30 seconds to simulate the sensation of stimulation, but then will immediately decrease and turn off. Stimulation intensity and duration were selected based on the most commonly used parameters in the literature.

Active/sham is set with a single toggle on our device and will be done in advance by a separate member of the research team. Participants will be blind to stimulation condition. Participants will be asked which tDCS condition they believed they were in on Day 2; in a previous study in our lab of 80 participants, participants were at chance in accurately identifying their condition (44/80 correctly identified their condition, with 22/40 sham and 22/40 active accurately identifying the condition).

Group assignment.

Based on random group assignment, subjects will complete the 35 minutes following informed consent as follows:

1. Active tDCS groups will receive active tDCS in one of the conditions outlined in section 2.1. for 20 minutes. The first 10 minutes will involve non-language tasks, and then the speech motor task will begin, and last approximately 25 minutes. The current will stop automatically after 20 minutes, and the speech motor learning task will continue.
2. Sham tDCS groups will receive sham tDCS, with the electrodes put on in one of the conditions outlined in section 2.1. The stimulation ramps up to 1mA over 30 seconds and then decreases and turns off. The behavioral tasks are identical to the active tDCS groups. The first 10 minutes will involve non-language tasks, and then the speech motor task will begin, and last approximately 25 minutes.

All participant groups will then engage in unrelated cognitive and linguistic tasks for 30 minutes, followed by short-term retention and generalization. All participants will return two days later for longer-term retention and generalization testing.

OUTCOME MEASURES

Cluster accuracy. All recorded productions containing consonant clusters will be transcribed using the acoustic waveform, spectrogram, and perception. The most common error type in producing these clusters is the insertion of a schwa vowel either between the two consonants (/gdivu/ -> [gEdivu]) or before the cluster (/gdivu/ -> [Egdivu]). Because these insertions are difficult for English speakers to perceive, we will use acoustic properties to identify the presence of a vowel. A vowel will be identified by the presence of formant structure in the spectrogram (particularly higher formants F2, F3, etc., as these are not confusable with f0) and a corresponding vocalic (periodic) portion in the acoustic waveform. Other errors such as consonant deletion (e.g., /gdivu/ -> [divu]) and substitution (e.g., /gdivu/ -> [glivu]) will be identified perceptually and verified with the acoustic record. The remaining sounds in the nonwords (e.g., the [ivu] portion of /gdivu/) will be transcribed perceptually. Cluster accuracy reflects the accuracy of the first two consonants only; whole nonword accuracy reflects the entire stimulus. For each participant, the scoring will be completed by a single coder who was blinded to the tDCS condition of the participant as well as the session that each token came from. Interrater reliability will evaluated in two ways. First, 25% of the participants will be coded completely by two separate individuals to compute point-to-point interrater agreement. Second, each /gd/ and /pt/ token from each speaker will be analyzed to determine if it contained epenthesis by two independent coders as they measure the duration of the burst-to-burst sequence.

Burst-to-burst duration. As a secondary measure of cluster acquisition, we will examine the duration from the stop burst of the first consonant to the stop burst of the second consonant in /gd/ and /pt/ initial words. We will include clusters produced accurately and with epenthesis. A decrease in this measure will reflect participants coming closer to the target articulation. The duration of vowels following the cluster will also be measured to include as a factor in our analyses as a proxy for speaking rate. Each /gd/ and /pt/ token will be scored by two independent coders for each of these measures, and they will also be coded for accuracy and error type. For each token where the measurements differed by more than 5 ms, two coders will re-examine the item to agree upon the measurement. These will be the final values used in the analyses. This process has been standardized in our lab in approaches to duration measures.

ELIGIBILITY:
Inclusion Criteria:

* native English speaker (learned English in the home from birth)
* no exposure to languages that contain the trained consonant clusters (e.g., Slavic languages, Greek, Hebrew).

Exclusion Criteria:

* a history of speech, language or hearing disorder
* not passing a hearing screening (40 dB HL; ANSI: 1983) at 500, 1000, 2000, 4000Hz binaurally
* presence of potential tDCS risk factors: damaged skin at site of stimulation; presence of electrically or magnetically activated implant (including pacemaker); and metal in any part of their body

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of accurately produced words from baseline to retention | Baseline, 2 days after training
  Measure will be taken from recordings during motor learning task and at two retention time points. Evaluation of accuracy of each word will be based upon the acoustic signal and the presence of incorrect sounds will be considered an error. Each word will be evaluated for accuracy, and the overall percentage will be the primary variable.

SECONDARY OUTCOMES:
Change in duration from first consonant to second consonant from baseline to retention | Baseline, 2 days after training
  We will use the acoustic record to measure the duration between the release burst of the first consonant to the release burst of the second consonant in words that begin with stop-stop consonant clusters (/pt/, /gd/). We use acoustic analysis software and identify the burst of each consonant based on acoustic landmarks.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Buchwald, PhD, Principal Investigator — New York University
Locations (1):
- New York University Department of Communicative Sciences and Disorders, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.